CLINICAL TRIAL: NCT07084454
Title: Geriatric Oncology Care in Brazil: Remote Geriatric Assessment-Driven Interventions With Supportive Care (The GAIN-S Trial in Brazil)
Brief Title: Geriatric Oncology Care in Brazil: Remote Geriatric Assessment-Driven Interventions With Supportive Care
Acronym: GAIN-S
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Cristiane Decat Bergerot, PhD (Other)
Collaborators: City of Hope Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Cristiane Decat Bergerot, PhD, Head of Supportive Care, Instituto Oncoclinicas
Organization: Instituto Oncoclinicas (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: InstitutoOncoclinicas; CCR-24-200 (Other Grant/Funding Number: Rising Tide Foundation for Clinical Cancer Research)
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Geriatric Assessment; Geriatric Oncology; Quality of Life; Functional Decline; Depression; Aging; Supportive Care in Cancer; Activities of Daily Living
Keywords: Geriatric Assessment; Geriatric Oncology; Older Adults with Cancer; Multidisciplinary Intervention; CARG-GA; Telehealth; Functional Status; Depression; Quality of Life; Brazil; Randomized Controlled Trial; Remote Care Delivery
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This is a multicenter, two-arm, parallel-group randomized controlled trial. Participants are randomized in a 1:1 ratio to receive either a telehealth-delivered, geriatric assessment-guided multidisciplinary intervention (GAIN-S) or standard of care. Randomization is stratified by institution and disease stage (stage I-III vs. IV), using variable block sizes.
Masking Description: This is an open-label trial because:
  * Participants know if they are receiving the GAIN-S intervention.
  * The care providers and multidisciplinary team also know which arm the participant is in.
  * Masking is not feasible due to the nature of the intervention (telehealth and tailored supportive care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GAIN-S Intervention Arm (Experimental): Participants in this arm will receive a telehealth-delivered, geriatric assessment (GA)-guided multidisciplinary supportive care intervention (GAIN-S). The intervention includes a comprehensive GA conducted remotely, with personalized recommendations reviewed by a multidisciplinary team (including oncologist, geriatrician, psychiatrist, psychologist, nutritionist, and fitness trainer). Patients will receive tailored supportive care consultations via telehealth, aiming to improve physical function, reduce depressive symptoms, and enhance quality of life during cancer treatment.
  Interventions: Other: GAIN-S Multidisciplinary Telehealth Intervention
- Standard of Care (SOC) Arm (Active Comparator): Participants in this arm will receive the usual oncology care provided by their treating physicians. They will complete the geriatric assessment (GA) before treatment initiation, and the results will be made available to their oncologist. Referrals to supportive care services will be made at the physician's discretion based on GA findings. Patients will receive standard follow-up and management without the structured, multidisciplinary telehealth intervention provided in the GAIN-S arm.
  Interventions: Other: Standard Oncology Care

INTERVENTIONS:
Other: GAIN-S Multidisciplinary Telehealth Intervention — This intervention delivers a comprehensive geriatric assessment (GA) via telehealth to older adults with cancer. Based on the GA results, a multidisciplinary team including oncologists, geriatricians, psychiatrists, psychologists, nutritionists, and certified fitness trainers provide personalized supportive care recommendations and consultations remotely. The goal is to improve physical function, reduce depressive symptoms, and enhance quality of life during cancer treatment.
  Other Names: GAIN-S; Geriatric Assessment-Guided Intervention; Telehealth GAIN
  Arms: GAIN-S Intervention Arm
Other: Standard Oncology Care — Participants receive the usual oncology care provided by their treating physicians without a structured geriatric assessment-driven intervention. Geriatric assessment results are shared with the treating oncologist, who may refer patients to supportive care services based on clinical judgment. No coordinated multidisciplinary telehealth intervention is provided.
  Other Names: Usual Care; SOC
  Arms: Standard of Care (SOC) Arm

SUMMARY:
The goal of this clinical trial is to determine whether a telehealth-delivered, geriatric assessment-guided supportive care program (GAIN-S) can improve health outcomes in older adults (age 65 and above) with solid tumors who are starting a new cancer treatment in Brazil. The main questions it aims to answer are:

* Does GAIN-S improve physical function, as measured by activities of daily living (ADL), after three months?
* Does GAIN-S reduce symptoms of depression and improve quality of life after three months?

Researchers will compare patients receiving the GAIN-S intervention to those receiving standard care to see if the intervention leads to better physical function, fewer symptoms of depression, and improved quality of life.

Participants will:

* Complete a geriatric assessment (CARG-GA) before and after treatment.
* Be randomized to either standard care or the GAIN-S intervention.
* If assigned to GAIN-S, receive tailored supportive care via telehealth, which may include consultations with a psychologist, psychiatrist, nutritionist, geriatrician, exercise physiologist, or other specialists based on their needs.

DETAILED DESCRIPTION:
This is a multicenter, randomized controlled trial evaluating the effectiveness of a telehealth-delivered, geriatric assessment-guided intervention (GAIN-S) in improving health outcomes for older adults with solid tumors who are initiating a new systemic cancer therapy (chemotherapy, immune checkpoint inhibitors, and/or tyrosine kinase inhibitors) in Brazil.

The intervention is adapted from the Geriatric Assessment and Intervention Network (GAIN) model and integrates multidisciplinary supportive care services delivered remotely. The study is conducted across 14 oncology practices, including both private and public institutions, located in the Midwest, South, Southwest, and North regions of Brazil.

A total of 350 participants aged 65 years and older will be enrolled and randomized 1:1 to either the GAIN-S intervention or standard of care (SOC). All participants will complete a validated geriatric assessment (CARG-GA) at baseline and again at 3 months. The CARG-GA evaluates functional status, comorbidities, psychological well-being, nutrition, cognitive status, social support, and fall risk.

In the intervention arm (GAIN-S), patients will receive a tailored set of supportive care services based on their GA results. The multidisciplinary team-consisting of a medical oncologist, geriatrician, psychologist, psychiatrist, nutritionist, and exercise physiologist-will review the GA findings and deliver recommendations via telehealth (e.g., video calls or phone). Patients may receive one or more remote consultations from team members depending on their individual needs.

In the SOC arm, GA results will be shared with the treating oncologist, but no structured intervention will be implemented unless a critical issue is identified (e.g., severe depression or cognitive impairment), in which case referrals may be made.

The primary outcome is change in physical function (Activities of Daily Living - ADL) from baseline to 3 months. Secondary outcomes include changes in depression symptoms (Geriatric Depression Scale - GDS) and health-related quality of life (FACT-G) from baseline to 3 months.

In addition to the main trial, a separate feasibility study will be conducted to evaluate the implementation of the GAIN-S intervention in public hospital settings. This feasibility study will recruit 50 patients from public hospitals in Brazil and will assess the practicality, acceptability, and potential barriers to delivering geriatric telehealth interventions in resource-limited environments.

The study aims to address key gaps in cancer care delivery for older adults in low- and middle-income countries, where access to geriatric-trained oncology professionals is limited. The use of telehealth and standardized GA tools seeks to provide a scalable model for personalized care and improve outcomes in this underserved population.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older at time of enrollment
* Diagnosed with a solid tumor cancer of any stage
* Scheduled to start a new systemic cancer therapy (chemotherapy, immune checkpoint inhibitors, and/or tyrosine kinase inhibitors)
* Able to provide written informed consent
* Physician approval for participation

Exclusion Criteria:

* Inability or unwillingness to comply with study procedures, including telehealth visits
* Cognitive or other impairments precluding participation as determined by the investigator
* Any condition that, in the investigator's opinion, would make the patient unsuitable for the study or interfere with study assessments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Function (Activities of Daily Living - ADL) Score | Baseline to 3 months after treatment initiation
  Physical function will be assessed by measuring changes in the Activities of Daily Living (ADL) score using the patient-reported portion of the CARG-GA. The primary objective is to determine if the GAIN-S intervention improves physical function compared to standard care.

SECONDARY OUTCOMES:
Change in Symptoms of Depression (Geriatric Depression Scale - GDS) | Baseline to 3 months after treatment initiation
  Depressive symptoms will be measured using the Geriatric Depression Scale (GDS). The study aims to evaluate whether the GAIN-S intervention reduces symptoms of depression compared to standard care.
Change in Health-Related Quality of Life (FACT-G Score) | Baseline to 3 months after treatment initiation
  Quality of life will be measured by the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire. The study will assess if the intervention stabilizes or improves quality of life compared to standard care.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Oncoclinicas, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding sharing individual participant data (IPD) is currently under consideration. Factors such as participant privacy, ethical approvals, and logistical aspects will be evaluated before a final plan is established. Updates on data sharing intentions will be provided as the study progresses.

REFERENCES:
- [Background] Mohile SG, Dale W, Somerfield MR, Schonberg MA, Boyd CM, Burhenn PS, Canin B, Cohen HJ, Holmes HM, Hopkins JO, Janelsins MC, Khorana AA, Klepin HD, Lichtman SM, Mustian KM, Tew WP, Hurria A. Practical Assessment and Management of Vulnerabilities in Older Patients Receiving Chemotherapy: ASCO Guideline for Geriatric Oncology. J Clin Oncol. 2018 Aug 1;36(22):2326-2347. doi: 10.1200/JCO.2018.78.8687. Epub 2018 May 21. PMID 29782209
- [Background] Dale W, Klepin HD, Williams GR, Alibhai SMH, Bergerot C, Brintzenhofeszoc K, Hopkins JO, Jhawer MP, Katheria V, Loh KP, Lowenstein LM, McKoy JM, Noronha V, Phillips T, Rosko AE, Ruegg T, Schiaffino MK, Simmons JF Jr, Subbiah I, Tew WP, Webb TL, Whitehead M, Somerfield MR, Mohile SG. Practical Assessment and Management of Vulnerabilities in Older Patients Receiving Systemic Cancer Therapy: ASCO Guideline Update. J Clin Oncol. 2023 Sep 10;41(26):4293-4312. doi: 10.1200/JCO.23.00933. Epub 2023 Jul 17. PMID 37459573
- [Background] Bergerot CD, Bergerot PG, Razavi M, Philip EJ, Lakhdari S, Franca MVDS, Molina LNM, Freitas ANS, Taveira MC, de Azeredo AC, Fuzita WH, Fernandes CM, Pio RB, de Araujo R, Couto MM, de Vasconcellos VF, Nonino MF, Lee D, de Matos Neto JN, Buso MM, Soto-Perez-de-Celis E, Dale W. Implementation and evaluation of a remote geriatric assessment and intervention program in Brazil. Cancer. 2023 Jul 1;129(13):2095-2102. doi: 10.1002/cncr.34759. Epub 2023 Mar 25. PMID 36964938
- [Background] Bergerot CD, Bergerot PG, Razavi M, Franca MVDS, da Silva JRG, Cerveira JA, Fuzita WH, de Azeredo AC, Dos Anjos GM, de Vasconcellos VF, Philip EJ, de Matos Neto JN, Canedo JF, Laloni MT, Ferreira CGM, Buso MM, Pal SK, Nipp R, El-Jawahri A, Soto-Perez-de-Celis E, Dale W. Telehealth Geriatric Assessment and Supportive Care Intervention (GAIN-S) Program: A Randomized Clinical Trial. J Natl Compr Canc Netw. 2025 Jun;23(6):219-226. doi: 10.6004/jnccn.2025.7020. PMID 40499588
- [Background] Soo WK, King MT, Pope A, Parente P, Darzins P, Davis ID. Integrated Geriatric Assessment and Treatment Effectiveness (INTEGERATE) in older people with cancer starting systemic anticancer treatment in Australia: a multicentre, open-label, randomised controlled trial. Lancet Healthy Longev. 2022 Sep;3(9):e617-e627. doi: 10.1016/S2666-7568(22)00169-6. Epub 2022 Aug 22. PMID 36102776
- [Background] Mohile SG, Mohamed MR, Xu H, Culakova E, Loh KP, Magnuson A, Flannery MA, Obrecht S, Gilmore N, Ramsdale E, Dunne RF, Wildes T, Plumb S, Patil A, Wells M, Lowenstein L, Janelsins M, Mustian K, Hopkins JO, Berenberg J, Anthony N, Dale W. Evaluation of geriatric assessment and management on the toxic effects of cancer treatment (GAP70+): a cluster-randomised study. Lancet. 2021 Nov 20;398(10314):1894-1904. doi: 10.1016/S0140-6736(21)01789-X. Epub 2021 Nov 3. PMID 34741815
- [Background] Li D, Sun CL, Kim H, Soto-Perez-de-Celis E, Chung V, Koczywas M, Fakih M, Chao J, Cabrera Chien L, Charles K, Hughes SFDS, Katheria V, Trent M, Roberts E, Jayani R, Moreno J, Kelly C, Sedrak MS, Dale W. Geriatric Assessment-Driven Intervention (GAIN) on Chemotherapy-Related Toxic Effects in Older Adults With Cancer: A Randomized Clinical Trial. JAMA Oncol. 2021 Nov 1;7(11):e214158. doi: 10.1001/jamaoncol.2021.4158. Epub 2021 Nov 18. PMID 34591080
- See also: This website provides a list of clinical trials currently being developed and conducted through the Cancer and Aging Research Group's Geriatric Oncology (CARG GOTO) program. — https://www.mycarg.org/?p=52053